CLINICAL TRIAL: NCT02995590
Title: Assessing Deformable Image Registration in the Lung Using Hyperpolarized-gas
Brief Title: Assessing Deformable Image Registration in the Lung Using Hyperpolarized-gas MRI
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Y. Michael Shim, MD, Associate Professor of Medicine, University of Virginia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 19112
Record Dates: First submitted 2016-12-13; First posted 2016-12-16 (Estimated); Last update posted 2020-11-04 (Actual); Status verified 2020-11

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MRI of lung motion during breathing (Experimental): * A medical history will be obtained defining any present and past history of respiratory illnesses, medications, and hospitalizations and the ability to have MR imaging.
  * A urine pregnancy test will be done for women of childbearing potential, who report the possibility that they might be pregnant.
  * Before and after MR imaging, a physical exam, spirometry, and a baseline %PO2 will be performed.
  * During the MR imaging procedure, the subject's heart rate and blood oxygen saturation will be monitored using an MR compatible pulse oximeter.
  * Once positioned in the MR scanner, conventional proton images of the thorax will be obtained to define the lung boundaries for subsequent image alignment. -Free breathing conventional MR imaging will be performed.
  * Hyperpolarized helium 3 imaging will be performed at breath hold.
  Interventions: Drug: Hyperpolarized He3

INTERVENTIONS:
Drug: Hyperpolarized He3 — Hyperpolarized Helium can be used as a Contrast Agent for Lung Images using MRI.
  Other Names: Helium study

SUMMARY:
Recently, the investigators have demonstrated a novel hyperpolarized helium tagging Magnetic Resonance Image (MRI) technique that is capable of directly, in vivo, and non-invasively measuring physiological lung deformation on a regional basis. This unique imaging technique holds great promise for assessing, validating, and improving the use of Deformable image Registration (DIR) algorithms in the lung. Our long term aim is to apply hyperpolarized gas tagging MRI to study lung biomechanics, develop more physiologically sound DIR algorithms for the lungs, and eventually improve radiotherapy of lung cancer. The overall aim of this application is to optimize the hyperpolarized helium tagging MRI technology and establish its usefulness for DIR assessment.

Our first objective is to develop and optimize a methodology based on 3 Dimensional (3D) hyperpolarized helium tagging MRI of healthy subjects, for directly measuring lung deformation between inhalation and exhalation. Our second objective is to develop physiologically sound digital thorax phantoms based on helium-3 tagging MRI of healthy subjects and demonstrate their use for DIR assessment in the lung. These phantoms will be used to evaluate a range different DIR algorithms, by comparing the errors between the DIR-derived deformation vector fields and the ground truth represented in the digital phantom. Successful completion of these aims will yield a novel methodology for DIR assessment in the lung for radiotherapy.

DETAILED DESCRIPTION:
The purpose of this study is to develop new ways to make medical images of the lungs and liver of adults using a technique called four-dimensional magnetic resonance imaging (4D-MRI). This technique produces three-dimensional movies of the inside of the chest and abdomen while the patient is breathing. (The fourth dimension is time!)

This new way of medical imaging is being developed to help cancer patients undergoing radiation therapy. Radiation therapy is used to treat cancerous tumors. For radiation therapy to be effective, the precise size, shape, and location of the tumor within the body must be known. A particular difficulty for radiation treatment of lung and liver cancer is that the tumor moves during treatment because the patient is breathing. Therefore, tumor motion must also be incorporated into the treatment plan. This study aims to improve radiation treatment planning through better targeting and dose estimation based on 4D-MRI. Before this new imaging method can be used for radiation treatment planning, it must be tested in living, breathing volunteers.

You are being asked to take part in a research study because you are a cancer patient or a healthy volunteer. You do not have to take part in this study. You should only agree to take part in this study after reading this consent form and discussing it with the study team. You may also discuss this with your family, friends, health care providers or others before you make a decision.

Though you may not be directly helped by being in this study, the information gained by doing this study may help others in the future. You might not want to take part in this study because of the temporary risk of discomfort during the time the subject is asked to lie still in the confined space of the MRI scanner. This discomfort may include claustrophobia (fear of being in a small space), feelings of warmth, muscle twitching due to excited nerves, and exposure to loud thumping noises produced by the MR scanner. If you are pregnant or think you may be pregnant, if would not be safe for you to be in this study.

ELIGIBILITY:
Inclusion Criteria:

* All subjects must be willing to participate and undergo the procedure, and be manageable as out-patients.
* Normal Subjects: Currently feeling well without respiratory symptoms.
* No history of lung disease.
* Never personally smoked (defined as less 100 cigarettes in their lifetime). -Secondhand smoke exposure is not an exclusion criterion.

Exclusion Criteria:

* Blood oxygen saturation of less than 92% as measured by pulse oximetry on the day of imaging.
* FEV1 percent predicted less than 80%.
* Pregnancy or lactation.
* Claustrophobia, inner ear implants, aneurysm or other surgical clips, metal foreign bodies in eye, pacemaker or other contraindication to MR scanning. Subjects with any implanted device that cannot be verified as MRI compliant will be excluded.
* Chest circumference greater than that of the xenon MR and/or helium coil. The circumference of the coil is approximately 42 inches.
* History of congenital cardiac disease, chronic renal failure, or cirrhosis.
* Inability to understand simple instructions or to hold still for approximately 10 seconds.
* History of respiratory infection within 2 weeks prior to the MR scan
* History of MI, stroke and/or poorly controlled hypertension.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Estimated)
Dates: Start 2016-07-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2021-12-15 (Estimated)

PRIMARY OUTCOMES:
Aim 1 | At time of MRI
  The difference between the deformation vector field derived from a given DIR algorithm (dDVF) and the known deformation vector field of the digital phantom (pDVF).

SECONDARY OUTCOMES:
Aim 2 | At time of MRI
  The Relationship between the DVF errors and motion amplitude.
Aim 3 | At time of MRI
  The relationship between the DVF and lung feature richness

CONTACTS AND LOCATIONS:
Overall Officials: Yun M Shim, MD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No